CLINICAL TRIAL: NCT04680390
Title: kINSHIP: Peer Navigators Addressing INtersectional Stigma to Improve HIV Prevention Among Criminal-justice Involved Women
Brief Title: HIV Prevention Peer Navigation for Justice Involved Women
Acronym: kINSHIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20-30358; R34DA050480 (NIH)
Record Dates: First submitted 2020-12-17; First posted 2020-12-23 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: HIV Infections; Stigma, Social
Keywords: Justice-involved population; Women's health; HIV prevention; Substance use; Intersectional stigma; Navigator
MeSH Terms: conditions — HIV Infections; Social Stigma; Substance-Related Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active-kINSHIP navigation intervention (Experimental): kINSHIP is a peer-led navigator intervention to address intersectional stigma and improve PrEP treatment initiation and engagement for justice-involved women. The key components of the kINSHIP intervention are to: 1) increase social support; 2) increase self-efficacy in accessing PrEP services; 3) enhance access to healthcare services; 4) improve adaptive coping skills to manage experiences of intersectional stigma.
  Interventions: Behavioral: Peer Navigators Addressing INtersectional Stigma to Improve HIV Prevention Among Criminal-Justice Involved Women
- Control-Standard Care (Active Comparator): The control arm will be standard-of-care, which is as-needed case management for justice-involved women.
  Interventions: Behavioral: Standard of care engagement practices

INTERVENTIONS:
Behavioral: Standard of care engagement practices — The control arm will be standard-of-care, which is as-needed case management for justice-involved women. The goals of case management services are to reduce recidivism, mitigate behavioral challenges, strengthen public safety, and build self-sufficiency skills. Case managers refer clients to appropriate services in the community (e.g., housing, food).
  Arms: Control-Standard Care
Behavioral: Peer Navigators Addressing INtersectional Stigma to Improve HIV Prevention Among Criminal-Justice Involved Women — kINSHIP is a peer-led navigator intervention to address intersectional stigma and improve PrEP treatment initiation and engagement for justice-involved women. The key components of the kINSHIP intervention are to: 1) increase social support; 2) increase self-efficacy in accessing PrEP services; 3) enhance access to healthcare services; 4) improve adaptive coping skills to manage experiences of intersectional stigma.
  Arms: Active-kINSHIP navigation intervention

SUMMARY:
Women involved in the criminal justice system have complex and highly stigmatized sexual and substance use risk profiles and are particularly vulnerable to, and experience, high rates of HIV. Criminal justice settings represent an important opportunity to address health disparities in HIV by linking women, who experience multiple, intersecting stigmas with innovative biomedical HIV prevention strategies, like pre-exposure prophylaxis (PrEP). The investigators propose to develop and test a peer-led patient navigation intervention for criminal-justice involved (CJI) women at risk of HIV acquisition to reduce intersectional stigma and improve uptake and linkage to PrEP services, thereby increasing access to PrEP and decreasing PrEP-related disparities.

DETAILED DESCRIPTION:
Stigma persists as a principal factor shaping HIV risk. Women involved in the criminal justice system have complex and highly stigmatized sexual and substance use risk profiles and are particularly vulnerable to, and experience, high rates of HIV. Pre-exposure prophylaxis, or PrEP, is an efficacious HIV prevention strategy, however, women at high-risk of HIV infection in the United States (US) are largely absent from national efforts to improve PrEP awareness and uptake. Criminal justice settings represent an important opportunity to address disparities in HIV by linking high-risk women, who experience multiple, intersecting stigmas with innovative biomedical HIV prevention strategies, like PrEP. Peer-led patient navigation interventions have demonstrated efficacy in building trust and reducing stigma and discrimination-related barriers to healthcare engagement, and hold strong potential to address multiple, intersecting stigmas and other multifactorial and complex barriers to PrEP acceptability, linkage, and uptake for criminal justice-involved women. The investigators propose to develop and test a peer-led patient navigator PrEP linkage intervention for women at risk for HIV acquisition who are on probation in San Francisco. Intervention development and study design will be guided by our team's pilot research, the Stigma and HIV Disparities Framework, and the PrEP Continuum of Care model. Study aims are to:1) Determine the content and structure of a peer-led PrEP screening and linkage navigation intervention (Project kINSHIP) for high-risk criminal justice-involved (CJI)-women; 2) Refine and test the content and structure of the kINSHIP intervention for CJI-women; and 3) Assess the feasibility, acceptability, and preliminary impact of the kINSHIP intervention on internalized stigma and the PrEP continuum of care in a pilot randomized trial. Formative qualitative work with key stakeholders, including women on probation, probation staff, and medical/public health staff in Aim1 will guide intervention development and testing in Aim 2. In Aim 3, the investigators will examine the primary outcome of PrEP service linkage and secondary outcomes such as time to linkage, PrEP prescription/initiation, and PrEP adherence/persistence. The investigators will explore how intersectional stigma may moderate intervention effects on linkage to PrEP. The proposed study has the potential to: 1) reduce the impact of intersectional stigma as a barrier to service care engagement, 2) inform PrEP care continuum estimates for criminal justice-involved women as well as identify barriers, and 3) create an intervention suitable for large-scale efficacy testing and translation to other criminal justice settings.

ELIGIBILITY:
Inclusion Criteria:

Women in San Francisco Adult Probation, ages 18-49 will be eligible if they:

* self-identify as HIV-negative;
* endorse risk behaviors in the past 6 months that call for consideration of PrEP per the Centers of Disease Control and Prevention risk indices;
* are English-Speaking.

Exclusion Criteria:

* Self-reported HIV infection;
* already on PrEP;
* observable cognitive/developmental delays or severe mental illness that would interfere with consent or participation.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2022-09-07 (Actual); Primary Completion 2024-11-06 (Actual); Study Completion 2024-11-06 (Actual)

PRIMARY OUTCOMES:
Linkage to PrEP services | 4 months post enrollment
  The primary outcome of PrEP linkage will be attendance at a PrEP services appointment, verified by medical records.

SECONDARY OUTCOMES:
Accepted PrEP referral | 4 months post enrollment
  Reported by the kINSHIP navigator.
Time to PrEP linkage | 4 months post enrollment
  Reported by the kINSHIP navigator and via medical record.
Accepted PrEP prescription | 4 months post enrollment
  Self-report and pharmacy collateral (if participant agrees).
PrEP initiation | 4 months post enrollment
  Self-report.
PrEP adherence | 4 months post enrollment
  Self-report.
PrEP persistence | 4 months post enrollment
  Self-report.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Dauria, PhD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No